CLINICAL TRIAL: NCT00227045
Title: The Iron Ion-Mycophenolate Mofetil Chelation Complex Interaction: A Two Phase Pharmacokinetic Study in Renal Allograft Recipients at the University of Michigan Transplant Program
Brief Title: CellCept/Iron Study: The Iron Ion-Mycophenolate Mofetil Chelation Complex Interaction in Renal Allograft Recipients
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Hoffmann-La Roche (Industry)
Other Study IDs: CEL305
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: End Stage Renal Disease
Keywords: Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The objective of this study is to determine the extent and magnitude of the pharmacokinetic drug interaction between mycophenolate mofetil (MFF) (under Css conditions) in the presence of iron in renal transplant recipients.

A two phase pharmacokinetic study will be conducted to determine the bioavailability of MMF (under steady state, Css, conditions) in the presence of two commonly prescribed iron formulations (polysaccharide iron complex and sustained release ferrous sulfate) in renal transplant recipients. This study will evaluate valuable clinical information to help better guide the appropriate utilization of the following formulations and dosing strategies:

1. Polysaccharide iron complex concomitant administration with MMF,
2. Sustained release ferrous sulfate concomitant administration with MMF,
3. Dose separation (2 hours) between MMF and iron (polysaccharide iron complex or sustained release [S.R.] ferrous sulfate)

DETAILED DESCRIPTION:
Following oral administration, MMF is rapidly absorbed and is presystemically hydrolyzed to its active form MPA in the liver. It is then metabolized by glucuronyl transferase to its inactive metabolite mycophenolic acid glucuronide (MPAG). MPA and MPAG also undergo a significant enterohepatic recirculation process, which is thought to contribute to the secondary peaks in the serum concentrations.

Pharmacokinetic studies in healthy volunteers have demonstrated the bioavailability to be ~94%. Previous studies have shown that many concomitantly administered medications including magnesium and aluminum containing antacids and cholestyramine, significantly impair bioavailability and decrease serum MPA AUCs from 37% and 40%, respectively.

However, of the potentially significant drug interactions involving MMF, iron may have the most clinically significant consequences. A large portion of the transplant population, particularly renal allograft recipients, experience anemia requiring iron supplementation. A single dose pharmacokinetic study conducted in seven healthy volunteers evaluated the effect of concomitant iron (delayed release preparation) administration on the absorption of MMF. This study reported a significant (89.7%) decrease in AUC among patients receiving concomitant iron and MMF. Although this study provides valuable information, it fails to address several clinically pertinent questions for transplant clinicians including:

1. the potential impact on steady state MPA kinetics in transplant patients,
2. effect of immediate release iron preparation compared with sustained release iron product, and
3. the effect of timing of the dose relative to administration of MMF.

ELIGIBILITY:
Inclusion Criteria:

* Patients prescribed iron and mycophenolate mofetil concomitantly
* The subject must be able to give informed consent for the study.
* Stable renal transplant patients age 18 years and older.
* At least 6 months status-post primary or secondary kidney transplant.
* Stable organ function
* Patients who have achieved therapeutic levels of cyclosporine, tacrolimus, or sirolimus.
* Patients on stable doses of cyclosporine, tacrolimus, or sirolimus. Defined as: No dosage adjustments within 2 weeks prior to study entry.
* Patients receiving ferrous sulfate iron preparations (either sustained release or immediate release preparations) or polysaccharide iron complex

Exclusion Criteria:

* Treated for acute rejection within the last 90 days
* Received other organ transplants in addition to kidney
* Pregnant or breast-feeding
* Use of iron supplements other than ferrous sulfate or polysaccharide iron complex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Park, PharmD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States